CLINICAL TRIAL: NCT03492671
Title: A Phase II Trial of Pre-operative Chemotherapy (With Gemcitabine and Nab- Paclitaxel) and Stereotactic Body Radiotherapy Followed by Surgery and Chemotherapy in Patients With Resectable Pancreatic Adenocarcinoma
Brief Title: Testing the Combination of Two Approved Chemotherapy Drugs and Radiation Prior to Surgery in Localized Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5170277
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pancreas Adenocarcinoma; Resectable Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Chemotherapy and SBRT (Experimental): Pre-Operative Chemotherapy: Within 28 days of study enrollment, subjects will receive a combination of Gemcitabine and Nab-paclitaxel for a maximum of four 28-day cycles. Gemcitabine 1000 mg/m2 IV on Days 1,8,15. Nab-paclitaxel 125 mg/m2 on Days 1,8,15.
  Post-Operative Chemotherapy: Within 5-10 weeks after surgery, subjects will receive a combination of Gemcitabine and Nab-paclitaxel for a maximum of two 28-day cycles. Gemcitabine 1000 mg/m2 IV on Days 1,8,15. Nab-paclitaxel 125 mg/m2 on Days 1,8,15.
  Standard Stereotactic Body Radiation Therapy (SBRT) fractionation of 6 Gy per day will be used for all patients to a total dose of 30 Gy.
  Interventions: Drug: Gemcitabine 1000 mg; Drug: nab-paclitaxel; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Gemcitabine 1000 mg — Pre-Operative: 1000 mg/m2 IV on days 1, 8, 15 (28 days cycles times 4 cycles) Post-Operative: 1000 mg/m2 IV on days 1, 8, 15 (28 days cycles times 2 cycles)
Drug: nab-paclitaxel — Pre-Operative: 125 mg/m2 IV on days 1, 8, 15 (28 days cycles times 4 cycles) Post-Operative: 125 mg/m2 IV on days 1, 8, 15 (28 days cycles times 2 cycles)
Radiation: Stereotactic Body Radiation Therapy — Standard Stereotactic Body Radiation Therapy (SBRT) fractionation of 6 Gy per day will be used for all patients to a total dose of 30 Gy.
  Other Names: SBRT

SUMMARY:
The purpose of this phase 2 research study is to determine whether a combination of chemotherapy drugs plus radiation therapy, given before surgery in resectable pancreactic cancer, can help to increase the chances of surgeons achieving and R0 resection. The chemotherapy drugs used are gemcitabine and nab-paclitaxel. These drugs are both approved by the FDA for use in treating adults with pancreatic adenocarcinoma. The investigational portion of this study is providing the chemotherapy drugs and radiation therapy before surgery. Primary Endpoint, R) resection rate ≥70%. Secondary Endpoints, Disease free survival, Overall survival , Perioperative mortality and morbidity.

DETAILED DESCRIPTION:
Primary Endpoint: R0 resection rate ≥ 70%

Secondary Endpoints: Disease free survival, Overall survival, Perioperative mortality and morbidity

Treatment should start within 28 days of registration. Pre-operative Chemotherapy Patients will receive a combination of the agents (gemcitabine and nab-paclitaxel) prior to surgery for a maximum of four cycles.

Gemcitabine 1000 mg-m2 IV on days 1, 8, 15 Nab-paclitaxel 125 mg-m2 IV on days 1, 8, 15 28 day cycles

Post-operative Chemotherapy Treatment should start within 5-10 weeks of surgery. Patients will receive a combination of the agents (gemcitabine and nab-paclitaxel) after surgery for maximum of two cycles.

Gemcitabine 1000 mg-m2 IV on days 1, 8, 15 Nab-paclitaxel 125 mg-m2 IV on days 1, 8, 15 28 day cycles

Radiation Therapy Immobilization and Treatment Planning CT Scan All patients will be immobilized in a full body immobilization device in the supine position.

A 4D-CT scan from T5 to L5-S1 with intravenous and oral contrast will be performed.

Radiation Toxicity All acute toxicities will be scored according to the NCI Common Toxicity Criteria v4.0. Late toxicity will be scored per RTOG guidelines.

Surgery, Pre-operative Re-staging Pre-operative evaluation should occur within 2-4 weeks prior to the planned surgery date. Based on the results of the pre-operative evaluation, the corresponding action below should be taken.

Radiological responding or stable disease: Patients should proceed to surgery per protocol.

Surgery Pancreatic resection should occur within 4-10 weeks after the last dose of preoperative chemotherapy or SBRT. Staging laparoscopy may be performed at the time of planned laparotomy but is not required.

Post-operative Restaging Evaluation should occur within 2 weeks prior to initiation of postoperative chemotherapy.

Tumor Response Evaluation (Adapted From RECIST 1.1) Assessment of overall tumor burden and measurable disease To assess objective response or future progression, it is necessary to estimate the overall tumor burden at baseline and use this as a comparator for subsequent measurements. Only patients with measurable disease at baseline should be included in protocols where objective tumor response is the primary endpoint. Measurable disease is defined by the presence of at least one measurable. In studies where the primary endpoint is tumor progression (either time to progression or proportion with progression at a fixed date), the protocol must specify if entry is restricted to those with measurable disease or whether patients having non-measurable disease only are also eligible.

ELIGIBILITY:
Inclusion Criteria (all criteria must apply):

* Cytologic or histologic proof of adenocarcinoma of the pancreas.
* Localized, potentially resectable tumors.
* Greater or equal to 18 years of age.
* ECOG performance status of 0 or 1.
* Adequate hematologic, renal and hepatic function as defined by:
* ANC greater or equal to 1,500 cells/mm3
* Platelets greater or equal to 100,000 cells/mm3
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Serum creatinine ≤ 2 x ULN • ALT ≤ 5 x ULN
* AST ≤ 5 x ULN
* No history of prior therapy for pancreatic cancer.
* No history of active infection requiring IV antibiotics at the start of study treatment
* Non-pregnant and non-breast-feeding.

Exclusion Criteria:

* Patient has borderline resectable or metastatic disease.
* History of malignancy in the last 5 years other than in situ cancer or basal or squamous cell skin cancer or malignancies cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years.
* Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Curative Intent Resection (R0) rate | Within 2 weeks prior to initiation of post-operative chemotherapy.
  Measure the rate of R0 resection with all margins microscopically clear.

SECONDARY OUTCOMES:
Disease Free Survival Rate | Every three months up to two years after resection.
  Subject will be followed post-resection for evidence of pancreatic cancer.
Overall Survival Rate | Every six months up to 6 years post-resection.
  Subject will be followed post-resection for overall survival rate.

CONTACTS AND LOCATIONS:
Overall Officials: Naveenraj Solomon, MD, Principal Investigator — Loma Linda University Cancer Center
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No